CLINICAL TRIAL: NCT04691323
Title: The Longitudinal Relationship of Hydroxyurea Adherence Behavior to Health-related Quality of Life, Barriers to Adherence and Habit Formation in Patients With Sickle Cell Disease.
Brief Title: The Longitudinal Relationship of HU Adherence to HRQOL, Barriers to Adherence and Habit in SCD.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sherif Badawy, MD, Assistant Professor, Department of Pediatrics, Division of Hematology, Oncology and Stem Cell Transplant, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 2020-3366; 1K23HL150232 (NIH)
Record Dates: First submitted 2020-12-24; First posted 2020-12-31 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease; Sickle B+ Thalassemia; Sickle Beta Zero Thalassemia; Sickle Cell Hemoglobin C
Keywords: sickle cell disease; hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HU-Go app intervention arm (Other): Participants will use the HU-Go app intervention arm for 12 months.
  Interventions: Other: HU-Go app

INTERVENTIONS:
Other: HU-Go app — A novel multifunctional mobile app (HU-Go) to improve adherence to hydroxyurea in patients with sickle cell disease

SUMMARY:
The primary objective of this study is to better understand factors contributing to variations in hydroxyurea (HU) adherence behavior in adolescents and young adults (AYA) with sickle cell disease (SCD). To meet this objective, the researchers will conduct a prospective cohort study to determine the longitudinal relationship between HU adherence and health-related quality of life (HRQOL) overtime among AYA with SCD. The long-term goal of this research is to promote medication adherence behavior and improve health outcomes in AYA with SCD.

DETAILED DESCRIPTION:
Sickle cell disease is the most common genetic disorder in the US, affecting about 100,000 Americans, and about 1 in 400 African American live births, incurring annual health care costs of $335 million. SCD can lead to serious complications including unpredictable, debilitating pain episodes, cardiopulmonary disease, stroke, and long-term end organ damage.These complications lead to significant declines in health-related quality of life (HRQOL) and other patient-reported outcomes (PROs), culminating in early mortality, particularly among AYA. Hydroxyurea, at present, is the main FDA approved medication for SCD that reduces morbidity and mortality, improves HRQoL and lowers healthcare utilization.However, adherence to HU remains suboptimal with only 35-50% of patients achieving high adherence (≥90%), particularly among AYA with SCD. Low HU adherence has been associated with worse health outcomes, poor HRQOL and increased healthcare utilization. Low HU adherence is multifactorial, especially in AYA with other competing priorities and vulnerability in developmental and psychological factors contributing to adherence behavior. The specific aim for this study is to determine the longitudinal relationship of HU adherence behavior to health-related quality of life, barriers to adherence and habit formation among AYA with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-21 years old
* Any sickle cell disease genotype
* On steady state of hydroxyurea for 2 months
* Own or have access to a smartphone
* Parents of patients that meet the eligibility criteria and are enrolled in the study will be included

Exclusion Criteria:

* Patients with recent hospitalizations within the past 7 days

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hydroxyurea adherence rate | 12 months
  Adherence rate is defined as number of given HU doses given, as captured by HU-Go app, divided by total number of doses expected during study period.

SECONDARY OUTCOMES:
Adherence to Hydroxyurea using PROMIS Medication Adherence Scale (PMAS) | 12 months
  Higher score indicating higher adherence to hydroxyurea
Adherence to Hydroxyurea using Visual Analogue Scale | 12 months
  Numerical value on a scale 0-100% (higher score indicating higher adherence to hydroxyurea)
Pain score using Patient reported outcomes measurement information system (PROMIS) measure | 12 months
  Patient reported outcomes measurement information system (PROMIS) measure for pain intensity, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points (higher T scores indicating worse pain).
Fatigue score using Patient reported outcomes measurement information system (PROMIS) measure | 12 months
  Patient reported outcomes measurement information system (PROMIS) measure for fatigue, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points (higher T scores indicating worse fatigue).
Physical function score using Patient reported outcomes measurement information system (PROMIS) measure | 12 months
  Patient reported outcomes measurement information system (PROMIS) measure for physical function, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points (lower T scores indicating worse physical function).
Depression score using Patient reported outcomes measurement information system (PROMIS) measure | 12 months
  Patient reported outcomes measurement information system (PROMIS) measure for depression, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points (higher T scores indicating worse depression).
Anxiety score using Patient reported outcomes measurement information system (PROMIS) measure | 12 months
  Patient reported outcomes measurement information system (PROMIS) measure for anxiety, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points (higher T scores indicating worse anxiety).
Peer relationships score using Patient reported outcomes measurement information system (PROMIS) measure | 12 months
  Patient reported outcomes measurement information system (PROMIS) measure for peer relationships, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points (lower T scores indicating worse peer relationships).
Codes and themes from qualitative data analysis | 12 months
  Semi-structured interviews focused on HU taking behavior, barriers to adherence and habit formation

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M. Badawy, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States